CLINICAL TRIAL: NCT03496376
Title: Effects of Thoracic Kinesio Taping on Pulmonary Functions, Respiratory Muscle Strength and Functional Capacity in COPD Patients
Brief Title: Effects of Thoracic Kinesio Taping on COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Murat TOMRUK, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1925-GOA
Record Dates: First submitted 2018-03-26; First posted 2018-04-12 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: COPD
Keywords: kinesio taping; COPD; functional capacity; pulmonary functions; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An assessor who was blinded to treatment groups assessed clinical outcomes before the treatment process. The same assessor was also repeated assessments at 6th week (at the end of treatment process)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping Group (Experimental): Kinesio Taping Group received three different deep breathing exercises (diaphragmatic, thoracic, and lateral basal), each consisting of three sets of 10 repetitions, with 30 seconds of rest between each set plus thoracic kinesio taping application.
  Interventions: Other: Kinesio Taping; Other: Deep Breathing Exercises
- Control Group (Active Comparator): Control Group received three different deep breathing exercises (diaphragmatic, thoracic, and lateral basal), each consisting of three sets of 10 repetitions, with 30 seconds of rest between each set.
  Interventions: Other: Deep Breathing Exercises

INTERVENTIONS:
Other: Kinesio Taping — The material used for thoracic kinesio taping application was Kinesio® Tex Gold™ (Kinesio Holding. Patients were instructed to sit upright on an armless chair with no back support, with knees flexed to 90 degrees, feet on the floor and arms relaxed. Kinesio tape was applied anteriorly and posteriorly to facilitate respiratory muscles (primarily diaphragm) along the subcostal area. Additionally, two more kinesio tapes were applied to upper trapezius and scalene muscles' area which lies between neck and acromion at both sides (left and right).
  Arms: Kinesio Taping Group
Other: Deep Breathing Exercises — Three different deep breathing exercises (diaphragmatic, thoracic, and lateral basal), each consisting of three sets of 10 repetitions, with 30 seconds of rest between each set.

SUMMARY:
The purpose of this study was to investigate the effect of kinseio taping on functional capacity, pulmonary functions, respiratory muscle strength, severity of dyspnea, severity of fatigue in Chronic Obstructive Pulmonary Disease (COPD). Assessment of patients was done baseline and 6th week.

Eligible patients for the study randomly allocated to Kinesio Taping Group (KTG), or Control Group (CG). Both groups received three different deep breathing exercises (diaphragmatic, thoracic, and lateral basal), each consisting of three sets of 10 repetitions, with 30 seconds of rest between each set. KTG also received thoracic kinesio taping application.

ELIGIBILITY:
Inclusion Criteria:

* aged 40 years and older,
* having stage II-III COPD diagnosis according to GOLD system and BODE Index by chest physician,
* unwilling to participate in any kind of pulmonary rehabilitation program for COPD,
* able to read, write, and understand Turkish; and
* willing and able to attend the study.

Exclusion Criteria:

* being in COPD exacerbation period,
* having neurological or musculoskeletal problems that would affect physical mobility,
* having unstable, severe heart disease(s) (heart failure, unstable hypertension, previous angina pectoris or myocardial infarction, heart valve problems),
* having scar, lesion or incision in the area of kinesio tape application,
* previous use of kinesio tape,
* having skin sensitivity against kinesio tape,
* malignancy,
* having mental and cognitive disorders that would affect cooperation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Change in functional capacity | Baseline, 6th week
  Six-minute walk test (6MWT) is a valid, reliable and useful test for assessing functional capacity of COPD patients. This test assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance.

SECONDARY OUTCOMES:
Change in pulmonary functions | Baseline, 6th week
  Pulmonary function test (PFT) is a generic term used to indicate a battery of studies or maneuvers that may be performed using standardized equipment to measure lung function.
Change in respiratory muscle strength | Baseline, 6th week
  Measurement of respiratory muscle strength is useful in order to detect respiratory muscle weakness and to quantify its severity. Respiratory muscle strength is assessed by mouth pressures sustained for 1 s during maximaş static manoeuvre against a closed shutter.
Change in severity of dyspnoea | Baseline, 6th week
  Modified Medical Research Council (mMRC) dyspnea scale is a valid and reliable test for measuring the severity of dyspnea of COPD patients. This scale ranges from 0 to 4. A higher value represents a worse outcome.
Change in severity of fatigue | Baseline, 6th week
  Modified Borg Scale (MBS) is a useful scale for severity of fatigue. This scale ranges from 0 to 10. A higher value represents a worse outcome (0=not at all, 10=maximal).

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül Üniversitesi School of Physical Therapy and Rehabilitation, Izmir, Turkey (Türkiye)